CLINICAL TRIAL: NCT07204132
Title: Clinical Application of a Novel Endoscopic Cryoablation Technique Combined With Immunotherapy (TECIC Model) in Bladder-Preserving Therapy for Bladder Cancer
Brief Title: Investigation Into the Integration of Intracavitary Cryoablation and Immunotherapy in Bladder-Preserving Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Shuxiong Zeng, associate chief physician, Changhai Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KTSB20250312016
Record Dates: First submitted 2025-09-17; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Bladder Cancer
Keywords: TECIC Model; Immunotherapy; Endoscopic Cryoablation Technique
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Based on patient preference, eligible subjects were assigned to the experimental group, which involv (Experimental): After successful administration of anesthesia, a transurethral resection cystoscope is used to perform transurethral bladder tumor resection (TURBT). Alternative methods such as laser resection can also be employed to remove the tumor as thoroughly as possible and obtain biopsy samples. Under the direct visualization of the resection scope, cryoablation is performed at the base of the tumor lesion. For a single lesion, at least two complete freezing-thawing cycles (defined as the freezing start of each cycle to the complete thawing end) are applied; the freezing duration of each cycle is 3 to 5 minutes. If the lesion is large, two additional freezing-thawing cycles can be applied in different areas of the lesion to ensure adequate coverage of the entire lesion area. Postoperatively, based on the pathological and immunohistochemical results, adjuvant immunotherapy is initiated.
  Interventions: Procedure: TURBT combined with cryoablation-assisted postoperative immunotherapy
- control group (Other): According to the guidelines, a radical cystectomy should be performed. At the same time, according to the specific situation, urinary diversion procedures such as bladder channeling, ileal bladder substitution, ureterocutaneous fistula, and in situ neobladder surgery (open, laparoscopic or robot-assisted) can be carried out. The biopsy and resected specimens should be sent for pathological examination. The postoperative adjuvant treatment plan is determined by the attending physician based on the patient's condition as appropriate.
  Interventions: Procedure: The conventional surgery treatment group

INTERVENTIONS:
Procedure: TURBT combined with cryoablation-assisted postoperative immunotherapy — After successful anesthesia, the patient underwent TURBT. Other methods such as laser resection could also be used. The tumor should be completely removed and biopsy specimens taken as much as possible. Then, under the direct vision of the electrocautery scope, cryoablation was performed on the base of the tumor lesion. The freezing area was single lesion and at least 2 freezing cycles were carried out (the freezing start to the rewarming end constituted one cycle), with each cycle lasting 3-5 minutes. If the lesion area was large, 2 more freezing cycles could be added at different positions of the lesion to ensure coverage of the lesion area. After the operation, based on the pathological and immunohistochemical results, adjuvant immunotherapy was initiated, and concurrent adjuvant rhythm chemotherapy was also combined.
  Arms: Based on patient preference, eligible subjects were assigned to the experimental group, which involv
Procedure: The conventional surgery treatment group — According to the guidelines, a radical cystectomy should be performed, and at the same time, a urinary diversion procedure should be carried out based on the specific situation, such as bladder channeling, ileal bladder substitution, ureterocutaneous fistula, in situ neobladder surgery, etc. (open, laparoscopic or robot-assisted methods are all acceptable). The biopsy and resected specimens should be sent for pathological examination. The postoperative adjuvant treatment plan is determined by the attending physician based on the patient's condition as appropriate.
  Arms: control group

SUMMARY:
Professional Translation:

This study is a single-center, prospective, non-randomized, parallel-controlled clinical trial initiated and conducted by the Department of Urology at the First Affiliated Hospital of Naval Medical University. The Principal Investigator is Professor Zhang Zhensheng, and the projected execution period for the project is from July 2025 to July 2027. The study aims to evaluate the efficacy and safety of an innovative integrated bladder-preserving treatment model-novel endoluminal precise cryoablation combined with Transurethral Resection of Bladder Tumor (TURBT), immunotherapy, and metronomic chemotherapy (the TECIC model)-in patients with high-risk non-muscle-invasive bladder cancer (NMIBC). Bladder cancer is a common malignant tumor of the urinary system. While radical cystectomy remains the standard therapy, it is associated with significant trauma, numerous complications, and substantially impacts patient quality of life. Existing bladder-preservation strategies, such as TURBT alone or trimodal therapy (chemoradiation), face challenges including high recurrence rates and variable efficacy. This research builds upon prior development and clinical exploration of a domestically developed novel endoluminal liquid nitrogen balloon cryoablation technology. This technology enables precise cryoablation of the tumor base under direct endoscopic vision, inducing immunogenic cell death, which theoretically can synergize with immunotherapy and chemotherapy, offering a new approach to bladder-preserving treatment.

The study plans to enroll 180 patients diagnosed with high-risk NMIBC via biopsy or TURBT. Patient preference will be a key factor in group assignment. The experimental group (n=90) will undergo TURBT combined with intraoperative endoluminal precise cryoablation (at least 2 freeze-thaw cycles per lesion, each cycle lasting 3-5 minutes), followed by adjuvant anti-PD-1 monoclonal antibody immunotherapy (e.g., Camrelizumab, Tislelizumab, etc., for at least 3-6 cycles) and metronomic chemotherapy with a Gemcitabine plus Cisplatin (GC) regimen (at least 4-6 cycles). The control group (n=90) will receive radical cystectomy and urinary diversion selected according to current guidelines and individual circumstances; postoperative adjuvant therapy will be at the discretion of the attending physician. The primary efficacy endpoint of the study is 5-year Overall Survival (OS). Secondary efficacy endpoints include the rate of local intravesical recurrence/progression, 1-year and 2-year OS, 1-year, 2-year, and 5-year Progression-Free Survival (PFS), as well as quality of life scores. The safety endpoint is the incidence of postoperative adverse events. Furthermore, the study will explore biomarkers such as changes in local immune infiltration (assessed by detecting multiple immune markers in biopsy tissue) and peripheral blood cytokine levels and immune cell function before and after treatment.

Statistical analysis will employ the Full Analysis Set (FAS), the Per Protocol Set (PPS), and a 1:1 propensity score matching analysis set to reduce selection bias. Analysis of the primary efficacy index will be conducted at a one-sided significance level of 0.025. In contrast, other indexes will use a two-sided significance level of 0.05, utilizing SAS 9.3 statistical software. Descriptive analysis, efficacy analysis, and safety analysis will be performed separately. This study will strictly adhere to the principles of the Declaration of Helsinki, relevant Chinese regulations, and Good Clinical Practice (GCP). The protocol has been submitted for review and approval by the Institutional Review Board (IRB)/Ethics Committee. All enrolled patients are required to provide written informed consent before participation. It is anticipated that this study will provide a new, effective, and minimally invasive treatment option that preserves bladder function and quality of life for patients with high-risk NMIBC, while also preliminarily investigating the mechanism of action of the TECIC model.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 85 years old, gender not restricted;
2. Clinically diagnosed as patients with bladder tumors, and classified as high-risk non-muscle-invasive bladder cancer through biopsy or TURBT staging.

   * High-risk non-muscle bladder cancer is defined as meeting any of the following criteria: ① T1 stage tumor; ② High-grade urothelial carcinoma; ③ Simultaneously meeting: multiple, recurrent and diameter > 3cm bladder cancer;
3. The number of tumors is no more than 5;
4. Have the intention to preserve the bladder;
5. Voluntarily sign the informed consent form and be able to cooperate throughout the trial.

Exclusion Criteria:

1. Preoperative imaging indicated involvement of organs around the bladder (such as ureters, prostate, rectum, etc.), the pelvic or abdominal wall, or lymph node metastasis (N1) and distant metastasis (M1) stage;
2. Preoperative imaging indicated hydronephrosis, pathology suggested carcinoma in situ or diagnostic TURBT indicated diffuse tumor growth during the procedure;
3. Known to be allergic to chemotherapy drugs and/or immunotherapy drugs;
4. Complicated with severe infectious diseases such as bacteremia and toxemia;
5. Complicated with severe coagulation dysfunction;
6. Suffering from serious diseases such as heart, brain, lung, liver, kidney, etc., and unable to tolerate surgery;
7. Suffering from other malignant tumors;
8. Pregnant or lactating women;
9. Complicated with severe complications such as urethral stenosis that cannot tolerate cystoscopy surgery;
10. Complicated with prohibited medications, including systemic anti-tumor drugs and immunosuppressants;
11. Participating in other clinical trials simultaneously;
12. Other situations that the investigator considers inappropriate for participating in this clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Five-year overall survival, OS | 24 months

SECONDARY OUTCOMES:
Local recurrence/progression rate within the bladder cavity | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- ChangHai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared publicly to ensure patient confidentiality and privacy, as the informed consent obtained from participants did not include provisions for public data sharing. Additionally, data sharing is restricted by institutional policies and national regulations governing personal information protection.